CLINICAL TRIAL: NCT00155948
Title: Estimation of Muscle Area and Thickness of Deep Cervical Muscle Contraction During Cervical and Limb Movements
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701132
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2004-04

CONDITIONS: Multifidus
Keywords: Ultrasonography; Cervical Multifidus

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to investigate the validity and reliability of measurement for cervical multifidus using ultrasonography, and to investigate cervical multifidus muscle function by the change pattern of multifidus thickness, and to compare the changes in muscle thickness among different resistance levels (rest, 25%, 50%, 75% and 100%) and different cervical levels (C4, C5 and C6).

DETAILED DESCRIPTION:
Cervical multifidus has specific sensory and motion function. However, it was unclear about muscle architectural change of cervical multifidus during head retraction manoeuvre with progressive resistance. The validity and reliability of measuring cervical multifidus using ultrasonography hasn't been proven.

In the pilot study, thickness, width and area of multifidus were measured at C4, C5 and C6 were measured using MRI and ultrasonography. The limit of agreement and the regression analysis were used to compare the results of two modalities. Besides, muscle thickness was repeatedly measured during the static and head retraction manoeuvre using ultrasonography by the same rater on the same day; the CVw and CVb were used to investigate reliability. In the main study, multifidus architecture measured in twenty asymptomatic subjects (24.3±4.7 yo, 5 women and 15 men) during head retraction manoeuvre with progressive resistance and during relaxation using ultrasonography apparatus with 10MHz linear transducer. ANOVA with repeated measurement and post-hoc analysis were to investigate the difference among different cervical levels and resistance force levels.

The results of the pilot study showed that the limit of agreement was ±0.20 cm and the moderate level of correlation (R2 ranged in 0.42~0.64) for muscle thickness measured between MRI and ultrasonography. For muscle thickness, the CVw values under static and under head retraction against maximum resistance were lower than 10%. In the main study, there was a curvilinear relationship between muscle thickness change and resistance, and the quadratic equations were the proper curves for estimation. There was significant difference of muscle thickness change within 50% of maximum retraction against resistance; and there was no significant difference among three cervical levels. It was suggested that muscle at C6 relaxed more slowly during the period from the beginning of relaxation.

In conclusion, the present study built a valid and reliable method for measuring continuous and dynamic changes of muscle thickness using ultrasonography. The results supported muscle function of cervical multifidus for segmental stability but not for force production.

ELIGIBILITY:
Inclusion Criteria:

* participants without posterior cervical pain within recent 3 months before entry the study

Exclusion Criteria:

* Posterior cervical pain
* Surgery over cervical spine

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2003-09; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-Fen Wang, Ph.D., Principal Investigator — School and graduate institute of Physical Therapy, National Taiwan University